CLINICAL TRIAL: NCT05093114
Title: Friends, Family and Food: Interactive Virtual Environments for Children With Food Allergies
Brief Title: Friends, Family & Food: Food Allergy App for Youth ( F3A-App )
Acronym: F3A-App
Status: Completed | Type: Observational
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: R42 HD075524 (Open Trial); R42HD075524 (NIH)
Record Dates: First submitted 2021-10-07; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-05

CONDITIONS: Food Allergy in Children
Keywords: Food Allergy; Intervention; Virtual; Pediatric
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Objective: This Phase II STTR grant incorporated user feedback collected in an earlier development project to build interactive, web-based software that helps children with food allergies learn about their condition and gain self-management skills. This highly interactive game allows children to progress through virtual scenes to help them learn about food avoidance, symptom detection, and reaction management. In addition, this project built gaming complexity, with more levels and game options, of the two interactive games "Label Learning: Like it or Lose it!" and "Reaction Action!".

DETAILED DESCRIPTION:
The central goal of this project was to develop an interactive, game-based application (App) for school-aged children (aged 8-12) with food allergies (FA) that would increase knowledge, improve behavioral skills for disease management, and ultimately reduce risk of negative outcomes. An effective FA intervention for children should target content areas of food avoidance and reaction management, and across these areas facilitate knowledge acquisition, develop behavioral skills, and provide practice using these skills in social contexts. Our Friends, Family, and Food App (F3A-App), consists of four related parts: (a) an interactive, game-based application that is the core of the program, (b) the experiential scenarios in interactive environments (e.g., school cafeteria vignette) that target knowledge and behavioral skills practice in social contexts, (c) two engaging multi-level games to build skills in food avoidance (Label Learning: Like it or Lose it!) and symptom assessment (Reaction Action!), and (d) a multi-tiered reward system that uses token economy-based reinforcement to enhance motivation and engagement (SeaLife Spectacular). From a user perspective, the interactive, game-based application provides opportunities to practice behavioral skills (e.g. negotiating pressures to accept trigger foods, requesting assistance from adults, responding to teasing/bullying) in role-play situations with immediate feedback and reinforcement.

In this Phase II project, we proposed to produce a fully-developed version of the F3A-App, including added content and enhanced features, and evaluate the final product in a randomized clinical trial.

The specific aims of Phase II were:

1. To refine the F3A-App based on the user feedback and data collected in Phase I.
2. To develop and field test additional content, including two additional interactive environments (family gathering, school pot-luck); and to increase gaming complexity (i.e. more levels and options) in Label Learning: Like it or Lose it! and Reaction Action! We conducted a small open trial in which 40 children with FA, ages 8-12, used selected segments containing the newly developed content. Children used the application for 2 weeks on their home computer or tablet. Feedback about device preference and usage was used to determine our focus in the Evaluation Stage (Aim 3).
3. To assess the efficacy of the F3A-App vs. Standard Care (brief office visit and educational handouts) in a randomized clinical trial with 100 children with FA, ages 8-12. We expected the F3A-App would improve children's FA knowledge and self-efficacy to manage FA (primary outcomes) and would increase parent-child communication regarding FA management relative to Standard Care (secondary outcome). Our crossover design also enabled us to evaluate combined effects of Standard Care and the F3A-App through typical treatment channels (e.g., is the greatest efficacy found after a physician refers family to use the App after an office visit?) This Phase II STTR targeted pediatric FA, a critical public health problem of increasing prevalence. Our approach was innovative by incorporating an emphasis on behavioral skills practice using a platform that is engaging, interactive, affordable, and has high potential for broad dissemination. We envision that the F3A-App will ultimately serve as a template for interactive, game-based applications for children with other chronic conditions requiring self-management, such as asthma, diabetes, and celiac disease.

This record describes only the Open Trial portion of this Phase II STTR project.

ELIGIBILITY:
Inclusion Criteria:

* child must be 8 -12 years of age
* child must have an active diagnosis of food allergy (FA), specifically one or more of the four most common FAs that may cause anaphylaxis (peanut, tree nut, milk, and egg), confirmed by a physician within the past two years
* child and parent must speak and read English
* child must have access to a computer with internet access
* child must have access to a smartphone or tablet

Exclusion Criteria:

* Any chronic health condition requiring substantial dietary self-management (e.g., diabetes).

Ages: 8 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: Children with food allergy to one of the four most common FAs that may cause anaphylaxis (peanut, tree nut, milk, and egg)
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2015-05-18 (Actual); Primary Completion 2016-02-02 (Actual); Study Completion 2016-02-02 (Actual)

PRIMARY OUTCOMES:
Feedback interviews | Session 2, about 5 weeks after Session 1 and post-intervention
  A semi-structured interview assessing child participants' opinions and feedback regarding game segments.

SECONDARY OUTCOMES:
Food Allergy Knowledge Questionnaire | Baseline (pre-intervention/control condition), and Follow up (post-intervention/control condition; approximately 5 week after baseline)
  Child report
Food Allergy Management Efficacy | Baseline (pre-intervention/control condition), and Follow up (post-intervention/control condition; approximately 5 week after baseline)
  Child report
Food Allergy Independent Measure | Baseline (pre-intervention/control condition), and Follow up (post-intervention/control condition; approximately 5 week after baseline)
  Parent/Caregiver report
Food Allergy Caregiver-Child Communication | Baseline (pre-intervention/control condition), and Follow up (post-intervention/control condition; approximately 5 week after baseline)
  Parent/Caregiver report

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Mann-Koepke, PhD, Study Chair — Eunice Kennedy Shriver National Institute of Child Health & Human Development (NICHD)

IPD SHARING:
Plan to Share IPD: No